CLINICAL TRIAL: NCT04199923
Title: Harnessing Muscle-specific Atrophy Susceptibility to Disentangle the Mechanisms of Disuse Atrophy in Human Skeletal Muscle Atrophy (iMOB)
Brief Title: Mechanisms of Disuse Atrophy in Human Skeletal Muscle (iMOB)
Acronym: iMOB
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Biotechnology and Biological Sciences Research Council (Other)
Responsible Party: Principal Investigator, Bethan Phillips, Professor of Translational Physiology, University of Nottingham
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1031809
Record Dates: First submitted 2019-11-26; First posted 2019-12-16 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Muscular Atrophy; Immobility Syndrome
MeSH Terms: conditions — Muscular Atrophy

STUDY DESIGN:
Intervention Model Description: unilateral limb immobilisation study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 15 Day immobilisation (Experimental): The dominant leg of young healthy patients (18-40 years without serious comorbidities) will be immobilised using a fixed knee brace and aircast boot for 15 continuous days
  Interventions: Behavioral: Single leg immobilisation
- 5 Day immobilisation young (Experimental): The dominant leg of young healthy patients (18-40 years without serious comorbidities) will be immobilised using a fixed knee brace and aircast boot for 5 continuous days
  Interventions: Behavioral: Single leg immobilisation
- 5 Day immobilisation old (Experimental): The dominant leg of aged patients (65-80 years without serious comorbidities) will be immobilised using a fixed knee brace and aircast boot for 5 continuous days
  Interventions: Behavioral: Single leg immobilisation

INTERVENTIONS:
Behavioral: Single leg immobilisation — Immobilisation with single leg suspension immobilisation

SUMMARY:
Loss of muscle can be caused by a variety of stimuli and results in reduced mobility and strength and also impacts whole body health. Whilst it is known that muscles waste the process by which this occurs is not well understood. Furthermore, whilst some muscles waste quickly others seem resistant to the effects of disuse.

This study aims to evaluate how quickly changes in muscles start to occur, and investigate the processes which underlie muscle atrophy. By studying muscles which waste quickly and those which are resistant to atrophy this study aims to identify the different processes which lead to muscle loss. This study will also evaluate the differences in muscle changes between young and old people.

DETAILED DESCRIPTION:
Skeletal muscles host ~40% of all protein in the body. Muscles are not only crucial for locomotion but also represent the body's largest metabolically active tissue, glucose disposal site and fuel reservoir for other organs in pathological conditions (i.e., supply of amino acids to the liver for gluconeogenesis). Muscle atrophy is characterized by a reduction in cross sectional area (CSA) and length and occurs in many common illnesses (e.g. cancers (1), renal/heart failure, sepsis, genetic diseases, neurodegenerative disorders etc). It is also prevalent in situations of reduced neural input such as leg casting after fractures (2), bed-rest, spinal cord injury (3), space flight and chronic physical inactivity. Atrophy results in a loss of muscle power and strength (which is related to increased morbidity and mortality (4)) and reduced capacities for whole-body glucose storage and metabolism which causes insulin resistance. Strategies to oppose atrophy are limited but include mechanical loading (5) and the synergistic anabolic effects of nutrients. Although muscle atrophy is of great clinical importance, relatively little mechanistic research has been done in humans. Thus, the aim of this study is to assess the link between the variation in muscle physiological responses to disuse atrophy with variation in protein turnover and molecular-networks. This will not only provide new hypotheses for physiological regulation of human muscle and generate 'intervention targets' derived from clinically relevant human studies, it will also improve understanding of whether the response to disuse is altered with age and determine if mechanistic differences in atrophy resistant and atrophy sensitive muscles might explain inter-muscular variation in susceptibility to atrophy.

This study aims to define the molecular and metabolic mechanisms causing disuse atrophy in both young and older individuals and explore how and why some muscles are protected against it. The study will also assess temporal aspects of disuse atrophy (in younger individuals only) to explore the mechanistic basis for the more rapid atrophy observed in the early days of disuse.

ELIGIBILITY:
Inclusion Criteria:

* Group 1 and 2: Male, Age 18-40, BMI 18-35
* Group 3: Male, Age 65-80, BMI 18-35

Exclusion Criteria:

* BMI > 35 / <18
* Female
* Personal or Family History of Venous Thromboembolism
* Significant medical comorbidities

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Changes in muscle volume (cm3) | 14 days in group 1. 5 days in groups 2 and 3
  MRI assessment of muscle volume in Tibialis Anterior (TA) and Medial Gastrocnemius (MG) in immobilised vs non-immobilised leg, pre and post immobilisation
Changes in muscle thickness (cm) | 14 days in group 1. 5 days in groups 2 and 3
  Ultrasound scan (USS) assessment of muscle thickness in Tibialis Anterior (TA) and Medial Gastrocnemius (MG) in immobilised vs non-immobilised leg, pre and post immobilisation
Changes in muscle cross surface area (cm2) | 14 days in group 1. 5 days in groups 2 and 3
  Ultrasound assessment of muscle cross surface area, in tibialis anterior (TA) and Medial Gastrocnemius (MG) in immobilised vs non-immobilised pre and post immobilisation
Changes in muscle fibre length (cm) | 14 days in group 1. 5 days in groups 2 and 3
  Ultrasound assessment of muscle fibre length in tibialis anterior (TA) and Medial Gastrocnemius (MG) in immobilised vs non-immobilised pre and post immobilisation
Changes in muscle fibre pennation angle (degrees) | 14 days in group 1. 5 days in groups 2 and 3
  Ultrasound assessment of muscle fibre pennation angle in tibialis anterior (TA) and Medial Gastrocnemius (MG) in immobilised vs non-immobilised pre and post immobilisation
Muscle Protein Synthesis (MPS) rate (%/hr) | Over 8 hours following immobilisation period
  IV tracer (Individual muscle MPS in TA+MG muscles in immobilised vs non immobilised legs)
Muscle Protein Breakdown (MPB) rate (%/hr) | Over 8 hours following immobilisation period
  IV Pulse tracers (IV tracers to give muscle specific MPB measures of TA+MG muscles in immobilised vs non-immobilised legs)

SECONDARY OUTCOMES:
Muscle blood flow | over 5 minutes (following immobilisation period)
  contrast enhanced ultrasound (CEUS) assessment of muscle blood flow in immobilised vs non-immobilised legs (TA+MG muscle specific)
Leg blood flow | Over 5 minutes (following immobilisation period)
  Doppler assessment of leg blood flow through common femoral artery in fed and fasted states in both immobilised and non-immobilised leg
Anabolic Signalling | 14 days in group 1. 5 days in groups 2 and 3
  Measurement of anabolic signalling pathways by western blot (comparison between immobilised vs non immobilised TA + MG muscles)
Catabolic Signaling | 14 days in group 1. 5 days in groups 2 and 3
  Measurement of proteasome and lysosomal and related catabolic signalling pathways by western blot (comparison between immobilised vs non immobilised TA + MG muscles)
RNA sequencing | 14 days in group 1. 5 days in groups 2 and 3
  complete RNA sequencing of immobilised vs non immobilised TA + MG muscles to determine gene set enrichment and pathway analysis
Histology | 14 days in group 1. 5 days in groups 2 and 3
  Morphological assessment of muscle fibres by histological techniques (comparing immobilised vs non immobilised TA + MG muscles)
Mitochondrial respiration | 14 days in group 1. 5 days in groups 2 and 3
  Measurement of mitochondrial respiration to assess different complex activity in immobilised vs non-immobilised TA + MG muscles
Intramuscular electromyography (iEMG) | 14 days in group 1. 5 days in groups 2 and 3
  Electrically induced maximum force development and fatigability in TA + MG muscles pre and post immobilisation
Muscle power | 14 days in group 1. 5 days in groups 2 and 3
  Assessment of changes in muscle power secondary to immobilisation through 1 rep max (kg) pre and post immobilisation
Cardio pulmonary fitness | 14 days in group 1. 5 days in groups 2 and 3
  Cardiopulmonary Exercise Testing (CPET) to assess changes in aerobic fitness (V02 max, anaerobic threshold and Watt Max) following immobilisation

CONTACTS AND LOCATIONS:
Overall Officials: Bethan E Phillips, PhD, Principal Investigator — University of Nottingham
Locations (1):
- Graduate Entry Medical School, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No